CLINICAL TRIAL: NCT05849337
Title: The Lóa Study: a Randomised Control Trial of a Brief Digital Intervention to Support Women Experiencing Intrusive Memories of Traumatic Events During Their Lifespan from the SAGA Cohort
Brief Title: The Lóa Study: a Brief Digital Intervention for Women with Intrusive Memories in the SAGA Cohort
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Arna Hauksdottir, Professor, University of Iceland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-186
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Intrusive Memories of Traumatic Event(s)
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Brief imagery-competing task (Experimental): Access to a brief imagery-competing task for 24 weeks (with optional researcher support during the study)
  Interventions: Behavioral: Brief imagery-competing task
- Brief psychoeducation and signposting task (Experimental): Access to psychoeducation and signposting regarding resources for psychological trauma in Iceland for 24 weeks (with optional researcher support during the study)
  Interventions: Behavioral: Brief psychoeducation and signposting task
- Treatment as usual (TAU) (Other): Routine care that participants would otherwise receive if having intrusive memories of traumatic events.
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Brief imagery-competing task — Two digital self-guided sessions of a brief digital imagery-competing task. A memory cue followed by playing a computer game with mental rotation instructions.
  Arms: Brief imagery-competing task
Behavioral: Brief psychoeducation and signposting task — Two digital self-guided sessions and access to psychoeducation and signposting regarding resources for psychological trauma in Iceland.
  Arms: Brief psychoeducation and signposting task
Other: Treatment as usual (TAU) — Routine care that participants would otherwise receive if having intrusive memories of traumatic events
  Arms: Treatment as usual (TAU)

SUMMARY:
Intrusive memories are sensory memories of a traumatic event(s) that spring to mind involuntarily, and can evoke strong emotions and disrupt functioning in daily life. Previous research has indicated that a brief cognitive intervention can prevent the development of intrusive memories as well as reduce the number of intrusive memories of long-standing trauma. Initial pilot work (using case studies and a pilot study, ClinicalTrials.gov identifier: NCT05089058) with women in Iceland indicates that the intervention is acceptable and feasible.

This randomised controlled trial will compare 3 arms to investigate if access to a cognitive task - either a brief self-guided imagery-competing task or a brief self-guided psychoeducation and signposting task - versus treatment as usual, can reduce the number of intrusive memories in week 5 (i.e., between-groups comparison), controlling for the number of intrusive memories in the baseline week.

The effect on the number of intrusive memories in week 5 (primary outcome), and other symptoms of post-traumatic stress, sleep and cognitive functioning will be tested.

This study is funded by the Icelandic Research Fund (11709-0270) and (200095-5601) and The Oak Foundation (OCAY-18-442).

DETAILED DESCRIPTION:
Participants will be recruited from the Stress and Gene Analysis (SAGA) Cohort, a population-based, longitudinal study of Icelandic women (www.afallasaga.is, see selected publications in the reference box below).

A statistical analysis plan will be prepared prior to the first interim analysis using both frequentist and Bayesian analyses for statistical inference.

Regular monitoring will be performed by Vistor to verify that the study is conducted, and data are generated, documented and reported in compliance with the protocol, good clinical practice (GCP) and the applicable regulatory guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Part of the SAGA cohort
* Aged 18 or above.
* Able to read, write and speak in Icelandic.
* Have internet access.
* Willing to be contacted remotely and having access to a smartphone or computer
* Experience 3 or more intrusive memories in the past week
* Willing to monitor intrusive memories in everyday life
* Willing and able to provide informed consent and complete study procedures
* Willing and able to be contacted by the research team during the study period.
* Have not taken part in a previous study of this intervention from this research team (e.g., the Loa case series, feasibility trial or pilot RCT).

Exclusion Criteria:

* Have fewer than three intrusive memories during the baseline week.
* Suicide risk in the initial assessment (response of 'nearly every day' to item 9 on PHQ-9).
* Those undergoing other treatments for post-traumatic stress disorder (PTSD) or its symptoms will not be excluded, so the study will be as inclusive as possible.

Ages: 18 Years to 73 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of intrusive memories of traumatic event(s) | Week 5 (all arms) controlling for run-in/baseline week
  The number of intrusive memories of traumatic events recorded by participants in a brief daily online intrusive memory diary for 7 days.

SECONDARY OUTCOMES:
Number of intrusive memories of the traumatic event(s) | Week 12 and week 24 follow-ups (all arms) controlling for run-in/baseline week
  The number of intrusive memories of traumatic events recorded by participants in a brief daily online intrusive memory diary for 7 days.
The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Baseline, week 5, week 12 and week 24 follow-ups
  A 20-item questionnaire assessing the severity of PTSD symptoms corresponding to the DSM-5 criteria for PTSD. Items are rated on a 5-point Likert scale ranging from 0 ("not at all") to 4 ("extremely"). Scores are summed to give a total severity score (ranging 0 to 80).
The Pittsburgh Sleep Quality Index Addendum for PTSD (PSQI-A) | Baseline, week 5, week 12 and week 24 follow-ups
  A 7-item questionnaire assessing the frequency of disruptive nocturnal behaviours (e.g., acting out dreams, episodes of terror or screaming). Respondents report symptoms over the past month on a 4-point Likert scale, ranging from 0 ("never in the past month") to 3 ("three or more times each week"). Total score ranges from 0 to 21 with higher scores indicating worse symptoms.
Cognitive Functions Scale | Baseline, week 5, week 12 and week 24 follow-ups
  An 11 item questionnaire about cognitive functions in particular memory and concentration. Items are rated on a 5-point scale, from 1 ("every day") to 5 ("never"). Total scores range from 11 to 55; higher scores indicate less concentration and memory difficulties.

OTHER OUTCOMES:
The Patient Health Questionnaire-9 (PHQ-9) | Baseline, week 5, week 12 and week 24 follow-ups
  A 9-item questionnaire assessing depression symptoms and their severity. Items are scored from 0 ( "not at all") to 3 ( "nearly every day"). The total score is the sum of all items and ranges from 0 to 27.
The Generalized Anxiety Disorder-7 scale (GAD-7) | Baseline, week 5, week 12 and week 24 follow-ups
  A 7-item questionnaire assessing severity of anxiety symptoms. Items are rated for how often they have bothered the respondent over the last two weeks, from 0 ("not at all") to 3 ("nearly every day"). The total score is the sum of all items and ranges from 0 to 21.
The Sheehan Disability Scale (SDS) | Baseline, week 5, week 12 and week 24 follow-ups
  A questionnaire assessing functional impairment across three domains: (1) Work/school, (2) social, and (3) family life. Domains are measured on an 11-point Likert scale, ranging from 0 ("not at all") to 10 ("extremely"). The scale is adapted to assess functional impairment associated with intrusive memories. The total score is the sum of all items and ranges from 0 to 30.
Quality of Life Scale (QOLS) | Baseline, week 5, week 12 and week 24 follow-ups
  16-item measure to assess quality of life on a 7-point Likert scale, ranging from 7 ("delighted") to 1 ("terrible"). The domains that are assessed are the following: (1) Social and community activities, (2) material and physical wellbeing, (3) relationships with other people, (4) personal development and fulfilment, and (5) recreation. The total score is the sum of all items and ranges from 16 to 112.
The World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Baseline, week 5, week 12 and week 24 follow-ups
  A 12-item questionnaire assessing difficulties due to health conditions, including mental or emotional problems (with reference to intrusive memories). Respondents rate how much difficulty they have had in each area in the past 30 days, from 0 ("none") to 4 ("extreme or cannot do"). The overall score is calculated as a percentage of the maximum possible score (i.e., 48 points). Lower scores indicate better functioning.
General Impact of intrusive memories | Baseline, week 5, week 12 and week 24 follow-ups
  2-items measuring the general impact of intrusive memories in terms of level of distress and vividness associated with the intrusions on a 11-point scale (ranging from 0 to 10), rated at the end of each diary week. High scores indicate higher levels of distress/vividness.
Acceptability and feasibility | Week 5
  Four questions to assess acceptability and feasibility of the both interventions. Rated on a 11-point scale (0 to 10) to measure the extent to which the individual would recommend the intervention and whether they consider it to be an acceptable way to reduce the frequency of intrusive memories. In addition, in this study, we include 1 item on the type of digital device used and 2 open-ended questions about the experience of using the digital platform.
Adverse events (AEs) | Week 5, week 12 and week 24 follow-ups
  A free-text response field measuring the occurrence of any health problems since the last contact.
Credibility/Expectancy Questionnaire | Right after randomization
  6-item questionnaire that rates to what degree the participant finds the intervention credible on a 11-point scale from 0 to 10. High scores indicate greater credibility.
Feedback Questionnaire | Week 5
  A 7-item questionnaire will assess participants' experience of using the intervention. The first five items assess how easy, helpful, distressing, burdensome and interesting participants found the intervention. This was assessed on a 11-point scale ranging from 0 ("not at all") to 10 ("very"). The last 2 free-text items ask how the brief cognitive task could be improved, and for any other comments.

CONTACTS AND LOCATIONS:
Overall Officials: Arna Hauksdóttir, PhD, Principal Investigator — University of Iceland; Emily Holmes, PhD, Principal Investigator — Uppsala University
Locations (1):
- University of Iceland, Sæmundargata 12, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: Yes
Anonymised research data will be made available on Open Science Framework (OSF) indefinitely
Supporting Information: Study Protocol, SAP
Time Frame: The aim is to share the Study Protocol and Statistical Analysis Plan upon the last participant completing the last visit. Supporting information mentioned above will be shared indefinitely and with no end date on the Open Science Framework (OSF) platform. The results of the study will be shared through open-access publications.
Access Criteria: Anonymised research data will be made available on Open Science Framework (OSF) indefinitely.
  OSF is an open-source web application that is freely accessible to the public and scientific community

REFERENCES:
- [Background] Jonsdottir SD, Hauksdottir A, Aspelund T, Jakobsdottir J, Runarsdottir H, Gudmundsdottir B, Tomasson G, Valdimarsdottir UA, Halldorsdottir T, Thordardottir EB. Risk factors for workplace sexual harassment and violence among a national cohort of women in Iceland: a cross-sectional study. Lancet Public Health. 2022 Sep;7(9):e763-e774. doi: 10.1016/S2468-2667(22)00201-8. PMID 36057275
- [Background] Yang Q, Thornorethardottir EB, Hauksdottir A, Aspelund T, Jakobsdottir J, Halldorsdottir T, Tomasson G, Runarsdottir H, Danielsdottir HB, Bertone-Johnson ER, Sjolander A, Fang F, Lu D, Valdimarsdottir UA. Association between adverse childhood experiences and premenstrual disorders: a cross-sectional analysis of 11,973 women. BMC Med. 2022 Feb 21;20(1):60. doi: 10.1186/s12916-022-02275-7. PMID 35184745
- [Background] Danielsdottir HB, Aspelund T, Thordardottir EB, Fall K, Fang F, Tomasson G, Runarsdottir H, Yang Q, Choi KW, Kennedy B, Halldorsdottir T, Lu D, Song H, Jakobsdottir J, Hauksdottir A, Valdimarsdottir UA. Adverse childhood experiences and resilience among adult women: A population-based study. Elife. 2022 Feb 1;11:e71770. doi: 10.7554/eLife.71770. PMID 35101173